CLINICAL TRIAL: NCT05556200
Title: A Phase II Trial of Camrelizumab in Combination With Apatinib for Neoadjuvant Treatment of Early-stage TNBC With a High Proportion of TILs
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Jieqiong Liu, M.D., Ph.D., Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NeoCAT
Record Dates: First submitted 2022-09-24; First posted 2022-09-27 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer; Triple-Negative Breast Cancer
Keywords: anti-PD-1 antibody; VEGFR2 TKI
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — spartalizumab; camrelizumab; apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experiment (Experimental): Eligible patients enrolled receive camrelizumab 200 mg, iv, d1, every 21 days (3 mg/kg if weight <50 kg) in combination with apatinib 250 mg, po, qd for neoadjuvant treatment for 8 cycles.
  Patients evaluated after neoadjuvant therapy with pCR receive 9 cycles of postoperative adjuvant camrelizumab (200 mg, iv, or 3 mg/kg if weight <50 kg, d1,q3W) + apatinib (250 mg, po, qd).
  Patients with non-pCR after neoadjuvant therapy receive adjuvant chemotherapy of the physician's choice (TPC).
  Interventions: Drug: Anti-PD-1 monoclonal antibody; Drug: VEGFR2 Tyrosine Kinase Inhibitor

INTERVENTIONS:
Drug: Anti-PD-1 monoclonal antibody — Camrelizumab 200 mg, iv, d1, q3W (3 mg/kg if weight <50 kg)
  Other Names: Camrelizumab
Drug: VEGFR2 Tyrosine Kinase Inhibitor — Apatinib 250 mg, po, qd
  Other Names: Apatinib

SUMMARY:
This is a phase II, open-labeled, multi-centered, single-arm, investigator-initiated clinical trial of camrelizumab (an anti-PD-1 antibody) in combination with apatinib (a VEGFR2 TKI) for neoadjuvant treatment of patients with triple-negative breast cancer and >10% tumor-infiltrating lymphocytes (TILs) in baseline breast tumors. We will enroll 58 subjects (Simon's two stage design). The study is designed to evaluate the efficacy and safety of camrelizumab in combination with apatinib in the neoadjuvant treatment of TNBC with a high proportion of TILs.

DETAILED DESCRIPTION:
This a phase II, open-labeled, multi-centered, single-arm, investigator-initiated clinical trial to assess the efficacy and safety of camrelizumab combination with apatinib in female patients age of 18 to 70 with TNBC, and baseline tumor-infiltrating lymphocytes > 10%. The number of patients to be included is 58 patients (Simon's two stage design). The primary objective is to assess the pCR. All enrolled patients will be treated with camrelizumab 200mg (iv. 3mg/kg for patient whose weight is below 50kg) on day 1 of each 21-day cycle, and apatinib 250mg daily (po, d1-d21).

ELIGIBILITY:
Inclusion Criteria:

1. Patients sign the written informed consent.
2. Women aged 18-70.
3. Patients with histologically confirmed operable invasive breast cancer (T1cN1-2 or T2-4N0-2)［ER-negative(IHC<1%), PR-negative(IHC<1%), HER2-negative（IHC-/+ or IHC++ and FISH/CISH-）］.
4. Percentage of tumor-infiltrating lymphocytes >10% in baseline breast tumor.
5. Patients with at least one measuring lesion that was conformed to RECIST v1.1 standard.
6. No previous breast cancer-related treatment, including chemotherapy, immunotherapy, endocrine therapy, radical surgery, or radiotherapy.
7. Patients can swallow pills.
8. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1.
9. Patients with a life expectancy of at least 12 weeks.
10. The patient's blood test results prior to enrollment met the following criteria： • Hb≥90g/L; • Plt≥100^9/L; • Serum albumin ≥3g/dL; • Neutrophils≥1.5^9/L;

    • TSH≤ normal upper limit (ULN);
    * ALT and AST ≤1.5 ULN (liver metastases ≤3 ULN);
    * TBIL ≤ULN (total bilirubin ≤1.5 ULN in Gilbert's syndrome or liver metastasis subjects);
    * ALT and AST ≤1.5 ULN (liver metastases ≤3 ULN);
    * AKP≤ 2.5 ULN;
    * Renal function within 7 days before the first administration: serum creatinine ≤1.5 ULN or creatinine clearance ≥60mL/min.
11. Female subjects of childbearing potential must have a negative serum pregnancy test within 7 days before the first dose and must be willing to use very efficient barrier methods of contraception for the course of the study through 6 months after the last dose of study treatment.

Exclusion Criteria:

1. Combination of other malignancies or previous malignancies other than breast cancer within the last 5 years, except for basal cell carcinoma or flat cell carcinoma of the skin or carcinoma in situ of the uterine cervix that has been adequately controlled by treatment.
2. Those who are not suitable for immunotherapy in combination with active infection.
3. The combination of severe non-malignant disease that would affect patient compliance or put the patient at risk.
4. Concomitant with other antineoplastic therapy or are participating in other clinical trials.
5. Male breast cancer, bilateral breast cancer or inflammatory breast cancer.
6. Patients with dementia, mental abnormality or any mental illness that prevents understanding of the informed consent form.
7. Patients with history of allergic reaction or contraindication to the use of any drug component of this trial.
8. Patients with any active autoimmune disease or a history of autoimmune disease (e.g., the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enterocolitis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism; subjects with vitiligo or whose asthma has completely resolved in childhood and does not require any intervention in adulthood may be included; (Patients with asthma that requires medical intervention with bronchodilators cannot be included).
9. Have cardiac clinical symptoms or disease that are not well controlled, such as:

(1) NYHA class 2 or higher heart failure; (2) Unstable angina pectoris; (3) Myocardial infarction within 1 year; (4) clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention.

10. Urine routine suggestive of urine protein ≥++, or confirmed 24-hour urine protein amount ≥1.0g.

11. Known presence of hereditary or acquired bleeding and thrombotic tendencies (e.g., hemophiliacs, coagulation disorders, thrombocytopenia, hypersplenism, etc.).

12. Patients with congenital or acquired immune deficiencies (e.g., HIV-infected individuals).

13. Live vaccines administered less than 4 weeks prior to study drug administration or possibly during the study.

14. Active tuberculosis. 15. Patients have received oral or intravenous antibiotic therapy within 2 weeks prior to neoadjuvant therapy.

16. Major surgical procedure within 4 weeks prior to the start of study treatment or anticipated need for major surgical procedure during the course of the study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Remission (pCR) rate | After neoadjuvant study treatment and surgery, up to approximately 24-26 weeks
  pCR rate (ypT0/Tis ypN0) is defined as the percentage of participants without residual invasive cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy by current American Joint Committee on Cancer (AJCC) staging criteria assessed by the local pathologist at the time of definitive surgery.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | After neoadjuvant study treatment and surgery, up to approximately 24-26 weeks
  The propotion of subjects with CR or PR according to RECIST v1.1.
Breast Conservation Rate | Up to approximately 24-26 weeks
  The percentage of patients who undergo breast-conserving surgery after neo-adjuvant therapy.
Incidence of Treatment-Emergent Adverse Events | From the first drug administration to within 90 days for the last dose
  Adverse events/serious adverse events.
Event-Free Survival (EFS) | Up to approximately 8 years
  Event-free survival (EFS) defined as the time from recruitment until documented disease recurrence, progression, or death from any cause in all participants. EFS events covered under "disease recurrence" will include local, regional, or distant recurrence and contralateral breast cancer. Ipsilateral or contralateral in situ disease and second primary non-breast cancers will not be counted as EFS events.
Overall Survival (OS) | Up to approximately 8 years
  defined as the time from randomization to death due to any cause.
Frequencies of Biomarkers | Up to approximately 24-26 weeks
  Biomarkers (including tumor/stromal PD-L1, stromal PD-1, tumor-infiltrating lymphocytes and tumor-infiltrating B cells, eg).

CONTACTS AND LOCATIONS:
Overall Officials: Jieqiong Liu, M.D., Ph.D., Principal Investigator — Sun Yet-sen Memorial Hospital
Locations (4):
- China (4):
  - Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - Shenshan Medical Center, Memorial Hospital of Sun Yat-sen University, Shanwei, Guangdong
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Second Military Medical University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided